CLINICAL TRIAL: NCT02807402
Title: Real World Evidence of the Effectiveness of Paritaprevir/r - Ombitasvir, + Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C - An Observational Study in Romania
Brief Title: Effectiveness of Paritaprevir/Ritonavir, Ombitasvir, + Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C in Romania
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Collaborators: IST GmbH, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-698
Record Dates: First submitted 2016-06-16; First posted 2016-06-21 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-08

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Paritaprevir; Ombitasvir; Dasabuvir; HCV
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin: Participants in this observational study received treatment with paritaprevir/ritonavir (r) and ombitasvir with or without dasabuvir ± ribavirin (RBV) for 12 or 24 weeks for the treatment of chronic hepatitis C (CHC), according to hepatitis C virus (HCV) genotype/subtype and stage of liver disease.
  The prescription of treatment regimen was at the discretion of the physician in accordance with local clinical practice and label, and was made independently from this observational study and preceded the decision to offer the patient the opportunity to participate in this study.

SUMMARY:
This study seeks to provide evidence of the effectiveness and obtain patient reported outcome (PRO) data for the interferon-free regimen of paritaprevir (PTV)/ritonavir (r) + ombitasvir (OBV), + dasabuvir (DSV), +/- ribavirin (RBV) in participants with chronic hepatitis C (CHC) in a real life setting across clinical practice patient populations in Romania.

ELIGIBILITY:
Inclusion Criteria:

Treatment-naïve or -experienced adult male or female patients with confirmed CHC, genotype 1, receiving combination therapy with the interferon-free paritaprevir/ritonavir and ombitasvir with dasabuvir ± RBV according to standard of care and in line with the current local label

If RBV is co-administered with the paritaprevir/ritonavir and ombitasvir with dasabuvir, it has been prescribed in line with the current local label (with special attention to contraception requirements and contraindication during pregnancy)

Patients must voluntarily sign and date a patient authorization to use and/or disclose his/her anonymized health data prior to inclusion into the study

Patient must not be participating or intending to participate in a concurrent interventional therapeutic trial

Exclusion Criteria:

None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical practice patient populations with chronic infection of HCV Genotype 1 (GT1)
Sampling Method: Non-Probability Sample
Enrollment: 522 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ferenci P, Bourgeois S, Buggisch P, Norris S, Curescu M, Larrey D, Marra F, Kleine H, Dorr P, Charafeddine M, Crown E, Bondin M, Back D, Flisiak R. Real-world safety and effectiveness of ombitasvir/paritaprevir/ritonavir +/- dasabuvir +/- ribavirin in hepatitis C virus genotype 1- and 4-infected patients with diverse comorbidities and comedications: A pooled analysis of post-marketing observational studies from 13 countries. J Viral Hepat. 2019 Jun;26(6):685-696. doi: 10.1111/jvh.13080. Epub 2019 Mar 5. PMID 30739368
- See also: Related Info — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this prospective, multi-center observational study a total of 522 adult patients chronically infected with hepatitis C virus (HCV) genotype 1 were enrolled by 22 centers in Romania.
Period: Overall Study
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Started | 522
Completed (HCV ribonucleic acid (RNA) treatment assessment performed at least 10 weeks post-treatment) | 516
Not Completed | 6
Not completed — Failure to Return | 1
Not completed — Death | 3
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 522
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (9.5)
Age, Customized [Count of Participants; unit: Participants]
  18-65 years | 374
  66-84 years | 147
  >=85 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 283
  Male | 239
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 522
Years Since Diagnosis of HCV Infection [Mean (Standard Deviation); unit: years] | 6.8 (5.69)
HCV Genotype [Count of Participants; unit: Participants]
  Genotype 1a | 4
  Genotype 1b | 517
  Genotype 1, Subtype Unknown | 1
Cirrhosis Status [Count of Participants; unit: Participants]
  No cirrhosis | 9
  Transition to cirrhosis | 32
  Cirrhosis | 481
HCV RNA [Median (Full Range); unit: log10 IU/mL] — Population: Enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype).
  log10 IU/mL
    number analyzed (Participants) | 519
    (all) | 5.87 [1.53 to 7.14]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virological Response 12 Weeks Post-treatment (SVR12)
Description: Sustained virologic response was defined as hepatitis C virus ribonucleic acid (HCV RNA) levels less than 50 IU/mL 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last dose of study drug (week 24 or 36 depending on the treatment regimen)
Population: Enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype). Three participants with genotype 1 prescribed paritaprevir/r and ombitasvir instead of paritaprevir/r, ombitasvir and dasabuvir (3DAA) were excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir ± Ribavirin: Participants in this observational study received treatment with paritaprevir/ritonavir (r) and ombitasvir with dasabuvir ± ribavirin (RBV) for 12 or 24 weeks for the treatment of chronic hepatitis C (CHC), according to hepatitis C virus (HCV) genotype/subtype and stage of liver disease.
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir ± Ribavirin
Number analyzed (Participants) | 519
percentage of participants | 98.1 [96.5 to 99.0]

2. Secondary Outcome: Percentage of Participants Achieving Virological Response at End of Treatment
Description: Virologic response was defined as hepatitis C virus ribonucleic acid (HCV RNA) levels less than 50 IU/mL.
Time Frame: End of treatment (week 12 or 24 depending on the treatment regimen)
Population: Enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir ± Ribavirin
Number analyzed (Participants) | 519
percentage of participants | 99.6 [98.6 to 99.9]

3. Secondary Outcome: Percentage of Participants in the Core Population With Sufficient Follow-up Data for SVR12 Who Achieved Sustained Virological Response 12 Weeks Post-treatment
Description: Sustained virologic response was defined as hepatitis C virus ribonucleic acid (HCV RNA) levels less than 50 IU/mL 12 weeks after the last dose of study drug.
  The core population with sufficient follow-up data regarding SVR12 included all core population participants who
  * had evaluable HCV RNA data ≥ 70 days after the last actual dose of paritaprevir/ritonavir, ombitasvir and dasabuvir
  * or a HCV RNA value ≥ 50 IU/mL at the last measurement post-baseline
  * or had HCV RNA < 50 IU/mL at the last measurement post-baseline, but no HCV RNA measurement ≥ 70 days after the last actual dose of paritaprevir/ritonavir, ombitasvir with dasabuvir due to reasons related to safety (e.g. dropped out due to adverse event) or virologic failure.
Time Frame: 12 weeks after the last dose of study drug (week 24 or 36 depending on the treatment regimen)
Population: Enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype), and with sufficient follow-up data regarding SVR12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir ± Ribavirin
Number analyzed (Participants) | 517
percentage of participants | 98.5 [97.0 to 99.2]

4. Secondary Outcome: Percentage of Participants With Relapse
Description: Relapse was defined as participants with a virologic response (VR; HCV RNA < 50 IU/mL) at end of treatment (EOT) followed by HCV RNA ≥ 50 IU/mL at any time after the end of treatment.
Time Frame: End of treatment (week 12 or 24 depending on the treatment regimen) and up to 24 weeks after the end of treatment.
Population: Enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics, and with VR at EOT and who completed treatment, and had ≥ 1 HCV RNA measurement ≥ 70 days post-treatment and were a treatment failure between EOT and post-treatment day 70.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir ± Ribavirin
Number analyzed (Participants) | 512
percentage of participants | 0.8 [0.3 to 2.0]

5. Secondary Outcome: Percentage of Participants With Breakthrough
Description: Breakthrough was defined as at least one documented HCV RNA < 50 IU/mL followed by HCV RNA ≥ 50 IU/mL during treatment.
Time Frame: 12 or 24 weeks (depending on the treatment regimen)
Population: Enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype) with virological response on-treatment and with at least one on-treatment measurement (including EOT) thereafter.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir ± Ribavirin
Number analyzed (Participants) | 36
percentage of participants | 0.00 [0.0 to 9.6]

6. Secondary Outcome: Percentage of Participants in Each Non-response Category 12 Weeks Post-treatment
Description: SVR12 non-response was categorized according to the following:
  * On-treatment virologic failure (breakthrough [at least one documented HCV RNA < 50 IU/mL followed by HCV RNA ≥ 50 IU/mL during treatment] or failure to suppress [each measured on-treatment HCV RNA value ≥ 50 IU/mL]);
  * Relapse, defined as HCV RNA < 50 IU/mL at EOT followed by HCV RNA ≥ 50 IU/mL post-treatment in patients who completed treatment (not more than 7 days shortened);
  * Death;
  * Premature treatment discontinuation with no on-treatment virological failure;
  * Missing SVR12 data and/or none of the above criteria.
Time Frame: 12 weeks after the last dose of study drug (week 24 or 36 depending on the treatment regimen)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir ± Ribavirin
Number analyzed (Participants) | 519
percentage of participants
  On-treatment virologic failure | 0.2
  Relapse | 0.8
  Death | 0.6
  Premature treatment discontinuation | 0.2
  None of the above criteria | 0.2

7. Secondary Outcome: Assigned Treatment Regimen
Description: Treatment regimen was assigned by the physician according to local practice and label. Participants could receive three direct-acting antiviral (DAA) drugs (paritaprevir/ritonavir, ombitasvir, and dasabuvir) with or without RBV for 12 or 24 weeks.
Time Frame: Baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir ± Ribavirin
Number analyzed (Participants) | 519
Participants
  3 DAA without RBV (12 weeks) | 73
  3 DAA + RBV (12 weeks) | 438
  3 DAA + RBV (24 weeks) | 8

8. Secondary Outcome: Percentage of the Direct Acting Antiviral (DAA) Dose Taken in Relation to the Target Dose of DAA
Description: Adherence to study treatment was calculated as:
  Cumulative dose taken / (initial prescribed dose * planned duration)
Time Frame: From first dose of study drug to end of treatment, 12 to 24 weeks depending on the treatment regimen.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir ± Ribavirin
Number analyzed (Participants) | 519
Participants
  > 105% | 6
  > 95% to ≤ 105% | 483
  > 80% to ≤ 95% | 28
  > 50% to ≤ 80% | 1
  ≤ 50% | 1

9. Secondary Outcome: Percentage of the Ribavirin Dose Taken in Relation to the Target Dose of Ribavirin
Description: Adherence to study treatment was calculated as:
  Cumulative dose taken / (initial prescribed dose * planned duration)
Time Frame: From first dose of study drug to end of treatment, 12 to 24 weeks depending on the treatment regimen
Population: Enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype), who were prescribed ribavirin, and with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir ± Ribavirin
Number analyzed (Participants) | 445
Participants
  > 105% | 6
  > 95% to ≤ 105% | 349
  > 80% to ≤ 95% | 39
  > 50% to ≤ 80% | 22
  ≤ 50% | 29

10. Secondary Outcome: Percentage of Ribavirin (RBV) Treatment Days in Relation to the Target Number of Ribavirin Treatment Days
Time Frame: From first dose of study drug to end of treatment, 12 to 24 weeks depending on the treatment regimen.
Population: Enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype), who were prescribed ribavirin.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir ± Ribavirin
Number analyzed (Participants) | 446
percentage of days | 94.5 (19.12)

11. Secondary Outcome: Number of Participants With Comorbidities
Time Frame: Baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin: Participants in this observational study received treatment with paritaprevir/ritonavir (r) and ombitasvir with or without dasabuvir ± ribavirin (RBV) for 12 or 24 weeks for the treatment of chronic hepatitis C (CHC), according to hepatitis C virus (HCV) genotype/subtype and stage of liver disease.
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 519
Participants
  Any comorbidity or coinfection | 335
  Any coinfection | 9
  Coinfection with human immunodeficiency virus (HIV | 4
  Coinfection with hepatitis B virus | 6

12. Secondary Outcome: Number of Participants Who Received Concomitant Medications
Description: Concomitant medication other than for chronic hepatitis C used from the time when the decision was made to initiate treatment with paritaprevir/ritonavir and ombitasvir with or without dasabuvir until after the last dose.
Time Frame: From first dose of study drug to end of treatment, 12 to 24 weeks depending on the treatment regimen
Population: Enrolled patients who received at least one dose of paritaprevir/ritonavir and ombitasvir with or without dasabuvir.
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 522
Participants | 263

13. Secondary Outcome: Change From Baseline in EuroQol 5 Dimension 5 Level (EQ-5D-5L) Index Score
Description: The EQ-5D-5L is a health state utility instrument that evaluates preference for health status. The 5 items in the EQ-5D-5L comprise 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which are rated on 5 levels of severity (1: indicating no problem, 2: indicating slight problems, 3: indicating moderate problems, 4: indicating severe problems, 5: indicating extreme problems), and a separate visual analog scale (VAS).
  Responses to the 5 dimension scores were combined and converted into a single preference-weighted health utility index score by applying country-specific weights.The range for EQ-5D-5L index score is 0 to 1 where '0' is defined as a health state equivalent to being dead and '1' is full health.The higher the score the better the health status.
Time Frame: Baseline, end of treatment (week 12 or 24 depending on the treatment regimen), and at 12 and 24 weeks after end of treatment
Population: Enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype) and with available data at baseline and each time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV: Participants received paritaprevir/ritonavir, ombitasvir, and dasabuvir without ribavirin for 12 weeks.
- Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV: Participants received paritaprevir/ritonavir, ombitasvir, and dasabuvir with ribavirin for 12 or 24 weeks.
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV
Number analyzed (Participants) | 55 | 319
units on a scale
  End of Treatment: number analyzed (Participants) | 51 | 294
  End of Treatment | 0.07 [0.04 to 0.10] | 0.04 [0.03 to 0.06]
  12 weeks post treatment: number analyzed (Participants) | 45 | 291
  12 weeks post treatment | 0.09 [0.06 to 0.13] | 0.08 [0.07 to 0.10]
  24 weeks post treatment: number analyzed (Participants) | 10 | 206
  24 weeks post treatment | 0.09 [0.01 to 0.16] | 0.10 [0.08 to 0.11]

14. Secondary Outcome: Change From Baseline in EuroQol 5 Dimension 5 Level (EQ-5D-5L) VAS Score
Description: The EQ-5D-5L is a health state utility instrument that evaluates preference for health status. with a separate visual analog scale (VAS).
  The VAS assesses overall health on a scale from 0 (worst health imaginable) to 100 (best health imaginable).
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV
Number analyzed (Participants) | 56 | 332
units on a scale
  End of Treatment: number analyzed (Participants) | 52 | 317
  End of Treatment | 10.9 [6.40 to 15.3] | 8.36 [6.55 to 10.2]
  12 weeks post treatment: number analyzed (Participants) | 47 | 305
  12 weeks post treatment | 13.9 [9.71 to 18.0] | 12.7 [11.1 to 14.4]
  24 weeks post treatment: number analyzed (Participants) | 10 | 220
  24 weeks post treatment | 18.8 [9.45 to 28.1] | 15.2 [13.2 to 17.2]

15. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Absenteeism
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Absenteeism indicates the percentage of work time missed due to health problems.
Time Frame: as for outcome 13
Population: Enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype). Participants who were employed with available data at baseline and each time point are included.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV
Number analyzed (Participants) | 10 | 67
percent impairment
  End of Treatment: number analyzed (Participants) | 6 | 47
  End of Treatment | -1.3 (3.1) | -1.4 (11.0)
  12 weeks post treatment: number analyzed (Participants) | 7 | 43
  12 weeks post treatment | -15.4 (37.4) | -3.8 (29.0)
  24 weeks post treatment: number analyzed (Participants) | 1 | 31
  24 weeks post treatment | -7.5 (NA) — Could not be calculated for one participant | -8.7 (34.4)

16. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Presenteeism
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Presenteeism indicates the percentage of impairment while working due to health problems.
Time Frame: as for outcome 13
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV
Number analyzed (Participants) | 9 | 68
percent impairment
  End of Treatment: number analyzed (Participants) | 6 | 54
  End of Treatment | -23.3 (29.4) | -8.5 (27.1)
  12 weeks post treatment: number analyzed (Participants) | 6 | 46
  12 weeks post treatment | -16.7 (30.1) | -10.4 (31.3)
  24 weeks post treatment: number analyzed (Participants) | 1 | 29
  24 weeks post treatment | -70.0 (NA) — Could not be calculated for one participant | -9.3 (21.4)

17. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Total Work Productivity Impairment (TWP)
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Total work productivity impairment (TWP) indicates the percentage of overall work impairment due to health problems.
Time Frame: as for outcome 13
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV
Number analyzed (Participants) | 10 | 63
percent impairment
  End of Treatment: number analyzed (Participants) | 5 | 44
  End of Treatment | -18.5 (30.5) | -8.7 (25.4)
  12 weeks post treatment: number analyzed (Participants) | 6 | 40
  12 weeks post treatment | -17.0 (30.6) | -11.5 (39.4)
  24 weeks post treatment: number analyzed (Participants) | 1 | 29
  24 weeks post treatment | -72.3 (NA) — Could not be calculated for one participant | -20.7 (31.4)

18. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Total Activity Impairment
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Total activity impairment (TAI) indicates the percentage of general (non-work) activity impairment due to health problems.
Time Frame: as for outcome 13
Population: Enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype) with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV
Number analyzed (Participants) | 54 | 320
percent impairment
  End of Treatment: number analyzed (Participants) | 49 | 282
  End of Treatment | -2.9 (29.7) | -10.4 (33.7)
  12 weeks post treatment: number analyzed (Participants) | 41 | 268
  12 weeks post treatment | -9.5 (31.0) | -10.5 (36.6)
  24 weeks post treatment: number analyzed (Participants) | 9 | 186
  24 weeks post treatment | -8.9 (49.9) | -11.5 (37.7)

19. Secondary Outcome: Change From Baseline in Patient Activation Measure 13 (PAM-13)
Description: PAM 13 is a measure used to assess the patient knowledge, skill, and confidence for self-management, consisting of 13 questions. Each of the 13 items can be answered with one of four possible response options, which are "disagree strongly" (1), "disagree" (2), "agree" (3), "agree strongly" (4). Scores were summed to calculate the overall raw score, then transformed to a scale with a theoretical range 0 to 100, based on calibration tables, with higher PAM scores indicating higher patient activation
Time Frame: Baseline and end of treatment (week 12 or 24 depending on the treatment regimen)
Population: Enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype) with available data at baseline and end of treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV
Number analyzed (Participants) | 29 | 184
units on a scale | -3.94 [-8.77 to 0.89] | -4.00 [-5.92 to -2.08]

20. Secondary Outcome: Change From Baseline in Beliefs Medication Questionnaire - (18-item BMQ)
Description: The BMQ consists of 2 sections and 18 questions to screen for patients' beliefs, attitudes and concerns about their medication. The BMQ-Specific section comprises two 5-item subscales assessing the necessity of and concerns about the prescribed medication (Specific-Necessity and Specific-Concerns). The BMQ-General section comprises two 4-item subscales assessing beliefs that medicines are harmful and overused by doctors in general (General-Harm and General-Overuse). The 18 items are rated on a Likert scale from 1 (strongly disagree) to 5 (strongly agree). Each subscale score ranges from 1 to 5. High scores in the Specific-Concerns scale represent the notion that adverse reactions are potentially harmful when taking medication on a regular basis, and high scores in the Specific-Necessity scale indicate the patient's need to adhere to medication to maintain health. High scores in the General-Harm and General-Overuse scales represent an overall negative perception of medication.
Time Frame: Baseline and end of treatment (week 12 or 24 depending on the treatment regimen)
Population: as for outcome 19
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV
Number analyzed (Participants) | 54 | 312
units on a scale
  Specific Concerns: number analyzed (Participants) | 51 | 287
  Specific Concerns | -0.26 [-0.49 to -0.03] | 0.06 [-0.03 to 0.16]
  Specific Necessity: number analyzed (Participants) | 51 | 299
  Specific Necessity | -0.07 [-0.26 to 0.12] | -0.21 [-0.28 to -0.13]
  General Overuse: number analyzed (Participants) | 51 | 295
  General Overuse | 0.01 [-0.20 to 0.23] | 0.01 [-0.08 to 0.10]
  General Harm: number analyzed (Participants) | 51 | 291
  General Harm | -0.02 [-0.21 to 0.18] | 0.10 [0.02 to 0.19]

21. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events, or Pregnancies
Time Frame: From first dose of study drug through 30 days after last dose (16 or 28 weeks depending on the treatment regimen). The over all median (minimum, maximum) duration of treatment was 84 (28, 175) days.
Population: All enrolled participants who received at least one dose of paritaprevir/ritonavir and ombitasvir with or without dasabuvir.
Measure: Count of Participants; unit: Participants
Groups:
- Paritaprevir/Ritonavir + Ombitasvir With RBV: Participants received paritaprevir/ritonavir and ombitasvir plus ribavirin for either 12 or 24 weeks.
- Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV: Participants received paritaprevir/ritonavir, ombitasvir, and dasabuvir without RBV for 12 weeks.
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir With RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV
Number analyzed (Participants) | 3 | 73 | 446
Participants
  Any adverse event | 0 | 6 | 82
  Serious adverse events | 0 | 3 | 17
  Pregnancies | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after last dose (16 or 28 weeks depending on the treatment regimen). The overall median (minimum, maximum) duration of treatment was 84 (28, 175) days.
Description: The safety population included all enrolled participants who received at least one dose of paritaprevir/ritonavir, ombitasvir, with or without dasabuvir.
Groups:
- Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With R+ RBV: Participants received paritaprevir/ritonavir, ombitasvir, and dasabuvir with ribavirin for 12 or 24 weeks.
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir With RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With R+ RBV
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/73 | 3/446
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/73 | 17/446
Other Adverse Events (participants affected / at risk) | 0/3 | 0/73 | 44/446
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paritaprevir/Ritonavir + Ombitasvir With RBV (N=3) | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV (N=73) | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With R+ RBV (N=446)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 6 (6)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTRIC VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
CHOLANGITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
JAUNDICE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 4 (4)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PYONEPHROSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paritaprevir/Ritonavir + Ombitasvir With RBV (N=3) | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV (N=73) | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With R+ RBV (N=446)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 44 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-03-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT02807402/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT02807402/SAP_001.pdf